CLINICAL TRIAL: NCT06677632
Title: Developing New Therapeutic Strategies to Counteract Synaptic and Cognitive Deficits in Alzheimer's Disease by Targeting zDHHC Enzymes
Brief Title: Targeting zDHHC Enzymes to Counteract Alzheimer's Disease
Acronym: zTARGETAD
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6858
Record Dates: First submitted 2024-07-31; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer's disease patients: TO DETERMINE THE EXPRESSION OF zDHHC ENZYMES AND CHANGES OF PROTEIN S- PALMITOYLATION IN THE hiPSC-DERIVED NEURONS AND BRAIN ORGANOIDS OBTAINED FROM AD PATIENTS
  Interventions: Other: Palmitoylation Enzyme Expression Profiling Study

INTERVENTIONS:
Other: Palmitoylation Enzyme Expression Profiling Study — The expression of 23 zDHHC enzymes will be studied in human post-mortem hippocampi of AD patients and controls that have already been collected from UK brain biobanks. zDHHC enzymes will be analyzed at both mRNA and protein levels by Real Time PCR and Western blotting techniques, respectively

SUMMARY:
Alzheimer's disease (AD) is a growing problem for aging populations worldwide and represents one of the most demanding challenges for biomedical and pharmacological research. All therapeutic attempts made so far based on current knowledge have proven scarcely effective, probably because the molecular mechanisms underlying the onset and progression of the disease remain poorly understood. Neuroinflammation and alteration of brain insulin signaling have been demonstrated to induce an AD-like phenotype and accelerate neurodegeneration in the hippocampus and neocortex of experimental models of AD. An increasing number of studies have shown the role of palmitoylated proteins in the regulation of synaptic plasticity and neuronal functions. Aberrant protein S-palmitoylation plays a pivotal role in brain insulin resistance (BIR)-dependent cognitive decline. Moreover, protein S-palmitoylation can target immune signaling pathways (e.g., STING, NOD1/2, JAK-STAT, T cell receptor signaling) and modulate inflammatory responses. Accordingly, S-palmitoylation has been shown to regulate localization and activity of several enzymes involved in cytokine receptor-mediated signaling and neuroinflammation.

Unpublished results showed aberrant protein S-palmitoylation in hippocampal tissues of both AD post-mortem brains and mouse experimental models of AD. Preliminary data reveal a key role of palmitoyltransferase enzymes (zDHHCs), which catalyze the S-palmitoylation of substrate proteins, in the development of neurodegeneration and cognitive deficits, suggesting that counteracting aberrant protein S-palmitoylation can be a novel therapeutic strategy for AD. Nevertheless, to date, therapeutic approaches targeting protein S-palmitoylation have not yet been attempted in AD and there are currently no available drugs specifically targeting zDHHCs.

The goal of this study is to develop novel therapeutic strategies targeting zDHHC enzymes to counteract S-palmitoylation-dependent synaptic and cognitive deficits in AD. Additionally, new biotechnological approaches aimed at inhibiting zDHHCs and their targets will be set up to expand the range of tools capable of interfering with altered protein S-palmitoylation in AD. To this end, a combination of different in vitro and in vivo techniques (electrophysiology, molecular biology, behavioral tests, microscopy studies) will be used in both animal and human models of AD, concurrent with innovative biotechnological strategies.

DETAILED DESCRIPTION:
S-palmitoylation is a protein post-translational modification involving the attachment of a palmitic acid molecule to cysteine residues. This modification influences protein trafficking toward cellular membranes and is finely regulated by a class of enzymes named zinc finger DHHC domain containing (zDHHC) S-acyltransferases. Proteins critically involved in Alzheimer's disease (AD), such as APP and BACE1, are targets of S-palmitoylation. Higher levels of S-palmitoylated proteins have been found in both post-mortem brain samples and brain organoids derived from induced pluripotent stem cells (hiPSCs) obtained from AD patients. Notably, both neurons and brain organoids derived from human AD hiPSCs exhibited molecular, morphological, and functional alterations reminiscent of AD. Intranasal administration of the palmitoylation inhibitor 2-bromopalmitate (2-BP) significantly counteracted LTP and memory deficits in 3×Tg-AD mice, extended lifespan, and decreased Aß deposition. Higher levels of zDHHC7 and zDHHC21 were also found in the hippocampus of 3×Tg-AD mice. Silencing of zDHHC7 in the hippocampus of 3×Tg-AD mice prevented cognitive deficits and Aß accumulation, along with counteracting palmitoylation of proteins critically involved in neuronal function. This confirms that modulation of zDHHC activity may be exploited for AD treatment.

The idea underlying this project is based on the assumption that zDHHC enzymes and alteration of protein S-palmitoylation play a key role in the onset and progression of AD. Dysregulated zDHHC activity and aberrant S-palmitoylation of neuronal proteins critically involved in the regulation of brain plasticity, neuroinflammation, and Aß metabolism can affect synaptic function, protein homeostasis, and mitochondrial activity, leading to the development of neurodegeneration and cognitive deficits. A druggable target, zDHHC7, has been identified to test the efficacy of novel therapeutic approaches. This study aims to validate a new strategy targeting zDHHC enzymes in human experimental models of AD. Human models will allow an understanding of the translation potential of these approaches to human disease, to be validated in subsequent clinical trials whose implementation exceeds the duration of the present project.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Age between 18 and 80 years
* Signed informed consent obtained

Exclusion Criteria:

* Patients suffering from other neurological diseases;
* Patients with coagulation disorders or in treatment with anticoagulant drugs;
* Patients suffering from dermatological diseases and connective tissue diseases;
* Patients suffering from other organic, psychiatric diseases or laboratory abnormalities could preclude participation or invalidate the study results;
* Inability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population will be drawn from adults receiving care at Clinica della Memoria at Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome, Italy
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Differences in zDHHC mRNA and protein expression levels between Alzheimer's disease (AD) models and control samples | Year 1
  Levels of zDHHC enzymes will be quantified in AD models and controls to measure potential differences. Real-Time PCR will be used to assess mRNA expression, while Western blotting will measure protein levels, providing detailed profiles of zDHHC expression.
Change in AD-associated deficits following zDHHC7 downregulation | Year 1
  Measurable changes in AD-associated deficits will be assessed after zDHHC7 downregulation, with a focus on alterations in cellular or molecular markers relevant to Alzheimer's pathology.

SECONDARY OUTCOMES:
Decrease in zDHHC enzyme expression in human experimental models of Alzheimer's disease | Year 2
  Levels of zDHHC enzyme expression will be measured to assess the impact of biotechnological interventions aimed at reducing zDHHC activity, with the goal of improving synaptic function in Alzheimer's disease models.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Grassi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy